CLINICAL TRIAL: NCT00564460
Title: On Label, Randomized, Double-Blind, Placebo-Controlled Trial of Preoperative Finasteride in Patients Undergoing Transurethral Resection of the Prostate (TURP)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Change of practice pattern. Green light laser
Sponsor: University of Alberta (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-2007; NCT00547430 (obsolete NCT alias)
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2009-11

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Finasteride 5 mg PO once daily for 8 weeks prior to TURP
  Interventions: Drug: Finasteride
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finasteride — Finasteride 5 mg PO once daily for 8 weeks prior to TURP
  Other Names: Proscar
  Arms: 1
Drug: Placebo — Placebo once daily for 8 weeks
  Arms: 2

SUMMARY:
Transurethral resection of the prostate (TURP) is a common treatment for benign prostatic hyperplasia (BPH). A common complication of TURP is blood loss. Preliminary data suggest that preoperative Finasteride, a 5 alpha-reductase inhibitor, may reduce blood loss during TURP. However, no study has examined the effect of preoperative Finasteride on clinical outcomes.

The study is a randomized, double-blind, placebo-controlled trial of preoperative Finasteride versus placebo in BPH patients undergoing TURP. Participants will be stratified by prostate volume (30 to 65 grams versus 66 to 100 grams) and randomly assigned to preoperative Finasteride or placebo. The primary end point is incidence of RBCT. Secondary end points are standard units of red blood cells transfused, variables related to perioperative bleeding (incidence of readmission, incidence of return to hospital, length of hospital stay), blood loss, change in serum hemoglobin, change in serum hematocrit, blood loss per gram of resected prostate tissue, operating time, change in AUA-SS, and change in HRQOL.

DETAILED DESCRIPTION:
The proposed trial is warranted for two main reasons. First, no study has examined the effect of preoperative Finasteride on important clinical outcomes such as the incidence of red blood cell transfusion, standard units of red blood cells transfused, readmission, return to hospital, and length of hospital stay. Second, a definitive randomized, double-blind, placebo-controlled trial documenting the efficacy of preoperative Finasteride on blood loss variables (e.g., intra-operative blood loss, change in serum hemoglobin) has yet to be conducted.

Participants will be recruited from the practices of Credentialed Urologists at the Alberta Urology Institute (AUI) and UAH in Edmonton, Alberta, Canada. The eligibility criteria include medical, demographic, and logistic criterion, and focus on internal validity as well as external validity. Eligibility criteria for the study are: (1) TRUS-confirmed prostate gland > 30 g, (2) 18 years of age or older, (3) fit and scheduled to receive TURP, (4) approval of the treating urologist, (5) able to understand and provide written informed consent in English, (6) no active psychiatric condition, (7) no previous Finasteride use, (8) normal DRE, (9) PSA greater than or equal to 4.0 ng/ml, (10) no current anticoagulation use (Heparin, Warfarin), (11) no ESRD, (12) no previous prostate or urethral surgery, and (13) not deemed to be a candidate for immediate surgery (within 1 week of initial evaluation).

ELIGIBILITY:
Inclusion Criteria:

1. TRUS-confirmed prostate gland > 30 g,
2. 18 years of age or older,
3. fit and scheduled to receive TURP,
4. approval of the treating urologist,
5. able to understand and provide written informed consent in English

   Exclusion Criteria:
6. active psychiatric condition,
7. previous Finasteride use,
8. abnormal DRE,
9. PSA greater than 4.0 ng/ml,
10. current anticoagulation use (Heparin, Warfarin),
11. ESRD,
12. previous prostate or urethral surgery,
13. deemed to be a candidate for immediate surgery (within 1 week of initial evaluation).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To compare the incidence of red blood cell transfusion after TURP in BPH patients randomized to receive preoperative Finasteride with those randomized to receive placebo. | During/post surgery

SECONDARY OUTCOMES:
To compare standard units of red blood cells transfused, variables related to perioperative bleeding, blood loss, serum hemoglobin, serum hematocrit, blood loss per gram of resected prostate tissue, operating time, AUA-SS, HRQOL after TURP | during/post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Howard Evans, MD, Principal Investigator — AUIRC/University of Alberta
Locations (1):
- Alberta Urology Institute, Edmonton, Alberta, Canada